CLINICAL TRIAL: NCT04469374
Title: The Effect of an Exercise Intervention for Preventing Osteoporosis Among Postmenopausal Women
Brief Title: Menopause Osteoporosis and Bone Intervention Using Lifestyle Exercise.
Acronym: MOBILE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Assessed for feasibility
Sponsor: Staffordshire University (Other)
Responsible Party: Principal Investigator, Jacky Forsyth, Associate Professor of Exercise Physiology, Staffordshire University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StaffsUni1
Record Dates: First submitted 2020-03-25; First posted 2020-07-14 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal

STUDY DESIGN:
Intervention Model Description: The project will be a randomised controlled trial, investigating between and within group differences pre- and post-intervention. There will be two trial arms: an intervention group and sham control group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will be blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Jumping exercise (Experimental): 10 rest-inserted jumps performed three times per week
  Interventions: Other: Jumping exercise
- Balance exercise (Sham Comparator): Single-leg balances for 60 seconds on each leg
  Interventions: Other: Balance exercise (sham control)

INTERVENTIONS:
Other: Jumping exercise — Participants will be required to perform 10 maximal vertical jumps, with a 10-s rest interval between each jump, using an arm swing in countermovement style on three days per week. The jumps will be performed without shoes on a hard surface. The jumps will be preceded by a warm-up lasting approximately 3 min and consisting of mobilisation exercises for the legs and lower back. Jumping will be progressed over time and in accordance with individual needs.
  Arms: Jumping exercise
Other: Balance exercise (sham control) — Participants will be required to perform balance exercises. Participants will be required to balance on one leg for up to 60 seconds (2 x 60 s is equivalent in duration to the 10 jumps). This exercise will be progressed.
  Arms: Balance exercise

SUMMARY:
Aim: to examine the effect of an exercise intervention for preventing osteoporosis among postmenopausal women.

Objectives:

To examine whether mean values for Broadband Ultrasound Attenuation (BUA) using Quantitative Ultrasound (QUS) among postmenopausal women following an eight-month exercise intervention (and at 3-month follow up), will be significantly higher than those obtained pre-intervention.

To examine whether mean BUA values among postmenopausal women following an eight-month exercise intervention (and at 3-month follow up) will be significantly higher than mean values obtained from participants in a control group undertaking sham exercises for an equivalent duration.

To examine the feasibility of the eight-month exercise intervention for a potential larger study (larger sample size, increased number of trial arms and increased outcome measures), in terms of recruitment, adherence, perceptions, barriers, and acceptability.

DETAILED DESCRIPTION:
Data will be collected at baseline, on study completion and at 3-month follow-up. Sequel to baseline data collection and ascertainment of eligibility, participants will be randomised into either the exercise intervention group or sham-control group. Randomisation will be through computer-generation of random numbers. Participants will be blinded to group allocation. Both groups will complete their required programme for eight months.

For the intervention group, participants will be required to perform 10 maximal vertical jumps, with a 10-s rest interval between each jump, using an arm swing in countermovement style on three days per week. The jumps will be performed without shoes on a hard surface. The jumps will be preceded by a warm-up lasting approximately 3 min and consisting of mobilisation exercises for the legs and lower back. Jumping will be progressed over time and in accordance with individual needs. Initially, jumping may be undertaken with the use of a handheld support (such as the back of a chair or table), should participants feel unstable. Jumps will be progressed to include multi-directional movements (jumping to the side, forwards, backwards, and diagonally). Natural progression will also occur as participants should improve their jump height with increased muscular explosiveness. Participants will be asked to fill out a simple, daily training log, stipulating when they have undertaken the exercise, in order for adherence to be assessed.

In the control group, participants will be required to perform balance exercises. The balancing exercises will be progressed and varied (to ensure adherence). Initially, the use of a handheld support (such as the back of the chair) can be used. Participants will be required to balance on one leg for up to 60 seconds (2 x 60 s is equivalent in duration to the 10 jumps). This exercise will initially be progressed using time, and then by doing the following: confounding the visual fixation (e.g., head turns), changing the centre of mass (e.g. arm/leg lifts); performing the stork balance (hands on hips, knee bent and supported by standing leg); reaching in multiple directions before regaining the initial stance; closing the eyes; reducing the base of support; and a combination of these activities. The starting level of difficulty will be prescribed by the researcher, according to each participant's functional ability. The balance exercises will be preceded by a warm-up lasting approximately 3 min and consisting of mobilisation exercises for the legs and lower back. The purpose of the sham exercise is to foster the perception of full participation in the study, in order to decrease attrition rates, and to blind participants to the intervention. The balance exercises, although not improving bone health, could decrease the risk of fracture, making the sham control group more ethical, owing to potential improvements, and limited risks.

To ensure quality control, digitised video clips of all exercises will be provided for the participants, who will be encouraged to perform the exercises as demonstrated on the video. The participants will be invited to one fully supervised group exercise session per month. These sessions will be used to monitor exercise quality, and to ensure progression is appropriate for each participant. Sessions will last 15-20 min. Attendance at these sessions will be monitored through registers. Apart from these supervised exercise sessions, participants will be given free choice to determine where and when they do the exercises. At the instructor-led session, training logs will be submitted. If they are unable to attend, participants will be asked to submit training logs electronically, or via post. To encourage adherence, an App will be used, which will enable weekly announcements to be posted, as well as emails and/or text reminders. Participants will be free to contact the researchers about any concerns they have during the intervention. Apart from the exercise undertaken, participants will be requested to maintain their usual exercise throughout the study.

To improve adherence, Bandura's Social Cognitive Theory for changing behaviour will be drawn upon. Specific constructs will include the knowledge and skills to perform the prescribed intervention, personal regulation of goal-directed health behaviour (self-control), and self-confidence in engaging in the exercise despite the absence of supervision. Reinforcement, i.e., activities that increase the propensity for adherence during the trial and beyond the study's lifespan, will also be addressed.

Participants' level of self-efficacy for engaging in lifestyle change will be assessed using a five-point Likert scale, from 'not at all confident' to 'very confident'. Participants will be asked to rate how confident they are to commit to engage in the exercise, irrespective of usual circumstances such as time constraints, stress, and fatigue. Assessment of self-efficacy will take place at the study onset, and at one-monthly intervals (via attendance at the supervised group sessions). With non-attendance, assessment will take place electronically. In the event of a low rating, modes of handling such situations without compromising commitment to the regime, will be given in relation to each participant's personal circumstances. In addition, at the study outset, participants will be asked to identify any circumstances that could motivate them to comply with the exercise, as well as any perceived barriers to adherence. Any issues will be discussed, and participants will be given the opportunity to design personalised adherence strategies. The aim will be to foster self-efficacy in both groups.

After the eight-month intervention, all females in the trial arm, who have completed the study, will be invited to take part in a focus group (in groups of 8, depending on numbers who volunteer for this), to examine participants' perceptions of the intervention. A topic guide will be used, which includes: An exploration of the perceived barriers to undertaking the exercise intervention; issues with adherence; acceptability of the intervention; adverse events; enjoyment; ratings of perceived exertion; how easily the intervention could be incorporated into lifestyle. At the end of the focus group, the topic guide will be checked to ensure that all areas had been covered. Focus groups will likely last between 45 and 60 min, although will continue until the researcher feels that data saturation has been reached. The focus groups will be audio-recorded and subsequently transcribed to facilitate analysis. Non-verbal participant behaviour will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

* postmenopausal; aged ≥50 years

Exclusion Criteria:

* Volunteers will be excluded from the study if they: are using any medicated that may affect bone turnover (e.g., corticosteroids, anticonvulsants, anticoagulants, calcitonin, bisphosphonates, raloxifene, denosumab and/or anabolic agents such as parathyroid hormone and growth hormone or steroids), including hormone replacement therapy and hormone-based contraception, within 6 months of starting the study; have or have had any bone, metabolic, kidney, liver, thyroid, gastro-intestinal or hormonal disorders or cancer, that may affect bone turnover; have a close family history of osteoporosis; have sustained a low trauma fragility fracture in the past 6 months; are a heavy smoking (>20 cigarettes/day); if they are already undertaking bone-specific jumping exercises or equivalent exercises; if they have an existing knee, hip or back injury or have any medical condition that would prevent them from completing the exercise. Additional exclusions at baseline testing will include: a low BUA score, i.e., estimated T score of <2.5; obesity as determined by body mass index of >35 km/m2, to minimise risk of strain or injury associated with the exercise. Participants will also not be able to undertake the bone scan if they have any foot swelling, as this can make results difficult to interpret.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
Broadband ultrasound attenuation | 8 months
  BUA as measured by Quantitative Ultrasound (UBIS 5000 Diagnostic Medical Systems, Montpellier, France).

SECONDARY OUTCOMES:
Timed up-and-go test | 8 months
  The test involves the participant starting in a seated position, walking 3 m, turning around, then walking back to the chair to sit down
Ground reaction force | 8 months
  To estimate the mechanical loading force due to the exercise, ground reaction force will be evaluated with the aid of a force plate (Advanced Mechanical Technology, Inc., AMTI).
Jump height | 8 months
  A countermovement jump test (with arms swinging naturally) will be used to assess change in jump height, using the Optojump system (Microgate S.r.l., Bolzano, Italy).
Questionnaire on quality of life | 8 months
  Quality of life using the Short-Form Health Survey, version 2; scoring from 0-100, with higher meaning better health

CONTACTS AND LOCATIONS:
Locations (1):
- Staffordshire University, Stoke, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No